CLINICAL TRIAL: NCT03396978
Title: The Influence of Gonadal Hormone Suppression on Adipocyte Lineage and the Microbiome
Acronym: BATE Plus
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator left the institution
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 17-1869
Record Dates: First submitted 2018-01-05; First posted 2018-01-11 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Adipose Tissue; Microbiome; Menopause

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GnRHag (Experimental): Participants will undergo 6 months of gonadotropin releasing hormone agonist (GnRHag) therapy (intramuscular injection of leuprolide acetate 3.75 mg for depot suspension; Lupron; TAP Pharmaceutical Products, Inc.; Lake Forest, IL) to chronically suppress ovarian hormones. A single injection of leuprolide acetate produces an initial stimulation (for up to 3 wk) followed by a prolonged suppression of pituitary gonadotropins and ovarian hormones. Repeated monthly dosing suppresses ovarian hormone secretion.
  Interventions: Other: GnRHag

INTERVENTIONS:
Other: GnRHag — Ovarian Hormone Suppression - the purpose of the intervention is not to study the drug, but the impact of the loss of ovarian hormones.

SUMMARY:
This research study plans to learn more about the role of female sex hormones on adipose tissue (or fat) and the gut microbiome (or the organisms that are in your digestive tract). The rationale for this study is that the rate at which women gain fat (especially in the stomach region) increases after menopause. It is thought to be due to the loss of estrogen because post-menopausal women who take estrogen gain less weight than those who do not take estrogen. Gut bacteria process estrogen and help determine the types of estrogen that circulate in the body. These bacteria can be changed with lifestyle factors such as diet, and may therefore, also affect the risk of diseases that are more common in women after menopause i.e., cardiovascular disease and cancer. In this study the investigators will obtain fat biopsies before and after 6 months of ovarian hormone suppression to measure how the fat cells change with the loss of female sex hormones (e.g., medical menopause). The investigators will also obtain stool and urine samples before and every month during the study to measure changes in the microbiome.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment into the parent protocol (COMIRB 16-1479 - The impact of estrogen status on the biological function of brown adipose tissue in women measured using quantitative PET/CT; PI - Edward Melanson, PhD)
* Participation in GnRHag intervention

Exclusion Criteria:

* Known allergy to lidocaine or other numbing medication
* Uncontrolled bleeding disorder or inability to withhold aspirin/NSAIDs or other blood thinning medications for 7 days prior to biopsy procedure.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Must be biological female. This study is investigating ovarian hormone suppression.
Enrollment: 5 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
Accumulation of Myeloid Cells | 8 months after enrollment of last participant
  Quantification of accumulation of myeloid cells in abdominal subcutaneous adipose tissue of women before and after gonadal hormone suppression as assessed by CD45+/CD14+ staining via flow cytometry of isolated adipose stroma.
Progenitor proliferation and adipogenic potential | 1 year after completion of last participant
  Progenitor proliferation measured by BrdU and adipogenic potential as measured by Oil Red-O staining with quantification by absorbance. Adipocyte specific gene/protein expression will be measured to confirm adipocyte status.
Gut microbial diversity | 1 year after completion of last participant
  Comparison of gut microbial diversity before and after gonadal hormone suppression at monthly intervals as assessed by sequencing of the V4 region of 16s rRNA

SECONDARY OUTCOMES:
In Vitro Metabolic Phenotyping | 2 years after completion of last participant
  in vitro measurement of lipid and glucose uptake, insulin and adrenergic sensitivity, and mitochondrial content.
β-glucuronidase activity | 2 years after completion of last participant
  analysis of β-glucuronidase activity in fecal samples from premenopausal women under gonadal hormone suppression therapy via a 96-well assay. This will serve as a direct measure of fecal capacity for estrogen metabolism.
Estrogen parent: metabolite ratios | 2 years after completion of last participant
  comparison of estrogen parent: metabolite ratios in relation to changes in bacterial diversity and enzyme activity. We will use UPLC-MS/MS metabolomics.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Gavin, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No